CLINICAL TRIAL: NCT01721005
Title: Screening Versus Routine Practice in Detection of Atrial Fibrillation in the Elderly Population of Lieto
Acronym: LietoAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: T31/2012
Record Dates: First submitted 2012-10-26; First posted 2012-11-02 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: atrial fibrillation; thromboembolism; patient education
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pulse palpation education (Other): The subject is educated to pulse palpation by registered cardiac nurse. The education time is limited to 10 minutes and done according preplanned education model
  Interventions: Other: Subject education to pulse palpation

INTERVENTIONS:
Other: Subject education to pulse palpation — The subject is educated to pulse palpation by registered cardiac nurse. The education time is limited to 10 minutes and done according preplanned education model.

SUMMARY:
The aim of this study is to evaluate the feasibility of patient education on feeling the own pulse irregularity in the elderly population of Lieto.

Prevalence of atrial fibrillation (AF) rises with age. Subjects have often symptoms like palpitation and discomfort but especially in elderly population there's significant quantity of persons who don't feel any symptoms and fail to seek for medical care for stroke prevention.

The main objectives in this study are to find out the prevalence of AF in the elderly population of Lieto, to assess the feasibility and reability of patient education on feeling one's pulse irregularity and the affect to the quality of life of the participating subjects and monitoring the possible increased burden to the public health care system.

The study contains two office visits with specified learning session and long-term phone-call follow-up.

DETAILED DESCRIPTION:
The main objectives in this study are to find out the prevalence of AF in the elderly population of Lieto, to assess the feasibility of patient education on feeling one's pulse irregularity and the affect to the quality of life of the participating subjects and monitoring the possible increased burden to the public health care system.

The study contains two office visits with specified learning session and long-term phone-call follow-up. A specially trained nurse will initially give a 10 min education on pulse palpation to each person and evaluate their capacity to learn pulse palpation. During followup visits the compliance of the patient and possible new arrhythmias plus quality of life issues are recorded and their ability of pulse palpation is evaluated by artificial hand where various kinds of pulses are transmitted.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 75 or over
* inhabitant of Lieto
* willing to participate

Exclusion Criteria:

* chronic atrial fibrillation
* ongoing anticoagulant treatment
* permanent institutional care

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-04; Primary Completion 2016-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The willingness to the pulse palpation and competence independently learn to feel own pulse. | 1 month control visit
  Based on learning session evaluated by nurse and objective evaluation of the learned skills by pulse-arm device and patient's pulse diary

SECONDARY OUTCOMES:
Number of patients with new atrial fibrillation detected during the study | At 1 year followup
  During the 1 year followup visit information on atrial fibrillation is gathered form the patients records and by interview

OTHER OUTCOMES:
Quality of life | 1 year followup visit
  EQ5D based evaluation
New atrial fibrillation at long-term followup | 5 year control
  Data on atrial fibrillation and thromboembolic complications is gathered from patient records and patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Juhani K Airaksinen, Professor, Principal Investigator — University of Turku
Locations (1):
- Härkätie community health center, Lieto, Finland

REFERENCES:
- [Derived] Jaakkola J, Virtanen R, Vasankari T, Salminen M, Airaksinen KEJ. Self-detection of atrial fibrillation in an aged population: three-year follow-up of the LietoAF intervention study. BMC Geriatr. 2017 Sep 16;17(1):218. doi: 10.1186/s12877-017-0607-0. PMID 28915862
- [Derived] Virtanen R, Kryssi V, Vasankari T, Salminen M, Kivela SL, Airaksinen KE. Self-detection of atrial fibrillation in an aged population: the LietoAF Study. Eur J Prev Cardiol. 2014 Nov;21(11):1437-42. doi: 10.1177/2047487313494041. Epub 2013 Jun 18. PMID 23780517